CLINICAL TRIAL: NCT06052787
Title: The Impact and Outcomes of Combined Cerebrolysin and Amantadine Sulfate Administration on Management of Patients With Traumatic Brain Injury in the ICU
Brief Title: Combined Cerebrolysin and Amantadine Sulfate Administration for Patients With Traumatic Brain Injury in the ICU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, ragab elshabasy, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: pharmacotherapy in TBI in ICU
Record Dates: First submitted 2023-09-19; First posted 2023-09-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — cerebrolysin; Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- standard of care (No Intervention): patients receiving the standard protocol of management of head injury in the ICU including
  * Ventilatory support, sedation and analgesia.
  * Hemodynamic support.
  * Hyperosmolar therapy.
  * Early post traumatic seizure prophylaxis.
  * Nutritional support: will try to start enteral feeds as soon as possible or total parenteral
  * nutrition will be used in the case of enteral feeding intolerance.
  * Temperature management: to maintain normothermia
  * Glycemic control: to maintain a glucose level of [140 -180 mg/dl]
  * Peptic ulcer prophylaxis:
  * Deep venous thrombosis (DVT) prophylaxis
- standard of care + Cerebrolysin (Experimental): patients receiving the standard protocol of management of head injury in the ICU plus 2 cycles of Cerebrolysin , each cycle 10 days, for total 20 days. From day 1 to day 10: cerebrolysin 50 ml once daily diluted in 250 ml normal saline intravenous infusion over 15 minutes. From day 21-30 : cerebrolysin 20 ml once daily diluted in 250 ml normal saline intravenous infusion over 15 minutes.
  Interventions: Drug: Cerebrolysin
- standard of care + Cerebrolysin + Amantadine sulfate (Experimental): patients receiving the standard protocol of management of head injury in the ICU plus amantadine sulfate at a dose of 100 mg twice daily on the day after randomization, with this dose will be continued for 14 days. The dose will be increased to 150 mg twice daily at week 3 and to 200 mg twice daily at week 4 (total 4 weeks), combined with 2 cycles of Cerebrolysin , each cycle 10 days, for total 20 days. From day 1 to day 10: cerebrolysin 50 ml once daily diluted in 250 ml normal saline intravenous infusion over 15 minutes. From day 21-30 : cerebrolysin 20 ml once daily diluted in 250 ml normal saline intravenous infusion over 15 minutes.
  Interventions: Drug: Cerebrolysin; Drug: amantadine sulfate

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin, a mixture of free amino acids and low molecular weight peptides, has a neurotrophic factor-like activity with immediate pleiotropic neuroprotective activity and long-term multimodal effects on endogenous post-lesional regulation. Cerebrolysin has been suggested to exert beneficial effects on neurobehavioural functions, cognitive performance , and neuro-motor recovery , as part of initial therapy in severe and moderate acute TBI.
  Arms: standard of care + Cerebrolysin; standard of care + Cerebrolysin + Amantadine sulfate
Drug: amantadine sulfate — The dopaminergic agonist amantadine enhances presynaptic dopamine release and inhibits dopamine reuptake, resulting in an increased amount of dopamine in the synaptic cleft. Amantadine may also increase the density of postsynaptic dopamine receptors and alter the conformation of these receptors. Amantadine acts as an NMDA receptor antagonist, blocking glutamate, an NMDA channel activator. This effect may be responsible for amantadine's possible beneficial effect soon after TBI
  Other Names: PK-MERZ
  Arms: standard of care + Cerebrolysin + Amantadine sulfate

SUMMARY:
The goal of this interventional study is to Measure the potential benefits of combined administration of cerebrolysin and amantadine sulfate as an add-on therapy to the standard management of patients admitted to the ICU with traumatic brain injury.

DETAILED DESCRIPTION:
Sixty-nine million individuals worldwide are estimated to sustain a TBI each year. The proportion of TBIs resulting from road traffic collisions was greatest in Africa and Southeast Asia (both 56%) and lowest in North America (25%).

Head injury remains the leading cause of death and severe disability in young adults, and it is also the most important single injury contributing to traumatic mortality and morbidity.

Traumatic brain injury (TBI) is a non-degenerative, non-congenital insult to the brain from an external mechanical force, possibly leading to permanent or temporary impairment of cognitive, physical, and psychosocial functions, with an associated diminished or altered state of consciousness.

There is growing evidence that medications may speed recovery by enhancing some neurological functions without impacting others. Pharmacotherapy is increasingly being used in both the sub-acute (less than 1 month post-TBI) and chronic (more than 1 month post-TBI) phases.

Amantadine is known to enhance neurotransmission, through the activation of dopamine-dependent brain circuits, and increases dopamine activity in pre-synapses and post- synapses, acting as an antagonist of the N-methyl D-aspartate receptor.

A study done on 184 patients of severe traumatic brain injury found better οutϲοme in the treatment group with amantadine sulfate as compared with the plaϲeƅο group over the 4-week treatment interval, and they demonstrated that amantadine improved recovery in patients with moderate and severe TBI.

Giaϲinο et al. used amantadine in 184 patients for 4 to 16 weeks after TBI, They found that Amantadine accelerated the pace of functional recovery during active treatment in patients with post-traumatic disorders of consciousness.

Cerebrolysin is a peptide preparation produced by a biotechnological process, a standardized enzymatic breakdown of purified, lipid-free brain proteins, a pharmacological agent with neuro-restorative and neuro-protective effects. It stimulates neuronal survival and differentiation, axonal growth and sprouting, the formation of new synapses, and neurogenesis in the dentate gyrus.

El Sayed et al. published a meta-analysis of the effect of different neuroprotective drugs in management of patients with traumatic brain injury resulting in substantial superiority of the cerebrolysin that was reflected in three-fold cognitive improvement and favorable Glasgow outcome score.

In a prospective, randomized, double-blind, placebo-controlled, parallel-group, multi-center phase IIIb/IV trial, the CAPTAIN I trial registered beneficial effects of Cerebrolysin after moderate to severe TBI.

The CAPTAIN II trial, enrolled 142 patients with moderate to severe TBI in a single-center, prospective, randomized, double-blind, placebo-controlled clinical trial confirms the benefits of Cerebrolysin in moderate to severe TBI.

In their retrospective case -control study, Lee et al., identified that an amantadine-plus-cerebrolysin regimen was shown to additively affect the conscious state of patients with prolonged disturbed consciousness secondary to acute brain injury, especially in patients who remained in a prolonged vegetative state.

* Type of the Study: a single-center, prospective, randomized, double-blinded (Patients, healthcare providers, data collectors, and outcome assessors are blinded to treatment allocation), and phase III clinical trial.
* Study setting: The study will be conducted at Ain Shams university hospitals.
* Study period: The study will be conducted over 18-24 months.
* Study population: patients admitted to the ICU with traumatic brain injury who are eligible according to the inclusion and exclusion criteria.

sample size : 150 patients in three groups , 50 patients in each group.

Study procedures:

All selected patients fulfilling the inclusion criteria will be subjected to the following on admission:

1. Formal written consent from patient relatives.
2. Clinical data of all patients will be recorded in the admission sheets of ICU, these data includes: Demographic characteristics, etiology of trauma ,GCS ,vital signs (mean arterial blood pressure (MAP), heart rate, oxygen saturation) ,electrocardiogram (ECG), Pupil (size, reactivity and if symmetrical or not) and any other body trauma as bone fractures, chest trauma ,etc.
3. The imaging findings: CT will be done to all patients on admission to ICU to detect the basal pathological lesions as brain edema, hemorrhagic contusions, extradural hemorrhage, and subdural hemorrhage.
4. The patients of the study will be randomly allocated into three groups.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years.
* Clinical diagnosis of head injury with moderate to severe TBI and a Glasgow coma scale (GCS) score of 7-12 at the time of hospital admission.
* Pre-hospital intubation/sedation/paralysis was accepted if the GCS score had been assessed before intubation/sedation/paralysis by trained staff.

Exclusion Criteria:

* History of intracranial interventions as well as ischemic or hemorrhagic stroke.
* Any neurological or non-neurological condition independent from TBI that might influence the functional outcome or other efficacy outcome measures.
* Clear clinical signs of intoxication influencing the evaluation, in the investigator's judgment.
* Patients with penetrating brain injury.
* Pregnancy or lactation.
* Patient with sever renal impairment (creatinine clearance > 30 ml/ minute).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
The Glasgow Coma Scale (GCS) | Glasgow coma scale (GCS) will be recorded on admission, and every week up to 6 weeks of trauma to detect the improvement in level of consciousness after management in all groups.
  The Glasgow Coma Scale (GCS) is used to assess the level of consciousness. It depends on the best motor, verbal and eye opening responses. GCS is used to classify insult severity as minor [GCS 13-15], moderate [GCS 9-12] and severe [GCS 3-8].
Disability rating-scale for severe head trauma (DRS) | DRS score will be collected at baseline and weekly through week 6 (during 4 weeks of treatment and 2 weeks after discontinuation).
  Disability rating-scale for severe head trauma (DRS) includes measures of arousability, awareness and responsivity of eye opening, verbalization, and motor response; cognitive ability of for Self Care Activities: understanding of feeding, dressing, and grooming; degree of assistance and supervision required; and employability. Scores range from 0 to 29, with higher values indicating greater disability.
Coma Recovery Scale-Revised (CRS-R) | CRS-R will be compared over the 4 weeks of treatment and during 2-weeks after discontinuation of treatment
  Coma Recovery Scale-Revised (CRS-R) is a standardized neurobehavioral assessment tool comprising six organized subscales (i.e., auditory, visual, motor, oro-motor,verbal, communication, and arousal); scores range from 0 to 23, with higher scores indicating a higher level of neurobehavioral function.
The Glasgow Outcome Scale (GOS) | atients in all groups will be assessed with The Glasgow Outcome Scale (GOS) on the end of 6th week.
  The Glasgow Outcome Scale (GOS) is one of the most widely used outcome instruments to assess global disability and recovery after traumatic brain injury. Patients in all groups will be assessed with The Glasgow Outcome Scale (GOS) on the end of 6th week which classify patients into: dead, vegetative state, severe disability, moderate disability and good recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab D Elshabasy, Principal Investigator — faculty of medicine - Ain shams university
Locations (1):
- Faculty of medicine - Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Sayed I, Zaki A, Fayed AM, Shehata GM, Abdelmonem S. A meta-analysis of the effect of different neuroprotective drugs in management of patients with traumatic brain injury. Neurosurg Rev. 2018 Apr;41(2):427-438. doi: 10.1007/s10143-016-0775-y. Epub 2016 Aug 18. PMID 27539610
- [Background] Chamoun RB, Robertson CS, Gopinath SP. Outcome in patients with blunt head trauma and a Glasgow Coma Scale score of 3 at presentation. J Neurosurg. 2009 Oct;111(4):683-7. doi: 10.3171/2009.2.JNS08817. PMID 19326973
- [Background] Dewan MC, Rattani A, Gupta S, Baticulon RE, Hung YC, Punchak M, Agrawal A, Adeleye AO, Shrime MG, Rubiano AM, Rosenfeld JV, Park KB. Estimating the global incidence of traumatic brain injury. J Neurosurg. 2018 Apr 27;130(4):1080-1097. doi: 10.3171/2017.10.JNS17352. Print 2019 Apr 1. PMID 29701556
- [Background] Giacino JT, Kalmar K, Whyte J. The JFK Coma Recovery Scale-Revised: measurement characteristics and diagnostic utility. Arch Phys Med Rehabil. 2004 Dec;85(12):2020-9. doi: 10.1016/j.apmr.2004.02.033. PMID 15605342
- [Background] Giacino JT, Whyte J, Bagiella E, Kalmar K, Childs N, Khademi A, Eifert B, Long D, Katz DI, Cho S, Yablon SA, Luther M, Hammond FM, Nordenbo A, Novak P, Mercer W, Maurer-Karattup P, Sherer M. Placebo-controlled trial of amantadine for severe traumatic brain injury. N Engl J Med. 2012 Mar 1;366(9):819-26. doi: 10.1056/NEJMoa1102609. PMID 22375973
- [Background] Gosseries O, Di H, Laureys S, Boly M. Measuring consciousness in severely damaged brains. Annu Rev Neurosci. 2014;37:457-78. doi: 10.1146/annurev-neuro-062012-170339. Epub 2014 Jun 23. PMID 25002279
- [Background] Jennett B, Bond M. Assessment of outcome after severe brain damage. Lancet. 1975 Mar 1;1(7905):480-4. doi: 10.1016/s0140-6736(75)92830-5. PMID 46957
- [Background] Lee S, Lee HH, Lee Y, Lee J. Additive effect of cerebrolysin and amantadine on disorders of consciousness secondary to acquired brain injury: A retrospective case-control study. J Rehabil Med. 2020 Feb 27;52(2):jrm00025. doi: 10.2340/16501977-2654. PMID 32057086
- [Background] Muresanu DF, Florian S, Homberg V, Matula C, von Steinbuchel N, Vos PE, von Wild K, Birle C, Muresanu I, Slavoaca D, Rosu OV, Strilciuc S, Vester J. Efficacy and safety of cerebrolysin in neurorecovery after moderate-severe traumatic brain injury: results from the CAPTAIN II trial. Neurol Sci. 2020 May;41(5):1171-1181. doi: 10.1007/s10072-019-04181-y. Epub 2020 Jan 2. PMID 31897941
- [Background] Obenaus A. (2022).Traumatic brain injury, Reference Module in Neuroscience and Biobehavioral Psychology, Elsevier.
- [Background] Poon W, Matula C, Vos PE, Muresanu DF, von Steinbuchel N, von Wild K, Homberg V, Wang E, Lee TMC, Strilciuc S, Vester JC. Safety and efficacy of Cerebrolysin in acute brain injury and neurorecovery: CAPTAIN I-a randomized, placebo-controlled, double-blind, Asian-Pacific trial. Neurol Sci. 2020 Feb;41(2):281-293. doi: 10.1007/s10072-019-04053-5. Epub 2019 Sep 7. PMID 31494820
- [Background] Rappaport M, Hall KM, Hopkins K, Belleza T, Cope DN. Disability rating scale for severe head trauma: coma to community. Arch Phys Med Rehabil. 1982 Mar;63(3):118-23. PMID 7073452
- [Background] Spritzer SD, Kinney CL, Condie J, Wellik KE, Hoffman-Snyder CR, Wingerchuk DM, Demaerschalk BM. Amantadine for patients with severe traumatic brain injury: a critically appraised topic. Neurologist. 2015 Jan;19(2):61-4. doi: 10.1097/NRL.0000000000000001. PMID 25607336
- [Background] Stan A, Birle C, Blesneag A, Iancu M. Cerebrolysin and early neurorehabilitation in patients with acute ischemic stroke: a prospective, randomized, placebo-controlled clinical study. J Med Life. 2017 Oct-Dec;10(4):216-222. PMID 29362596
- [Background] Talsky A, Laura R. Pacione, Tammy Shaw, Lori Wasserman, Adam Lenny, Amol Verma, Gillian Hurwitz, Robyn Waxman, Andrew Morgan, Shree Bhalerao .(2011).Pharmacological interventions for traumatic brain injury. BC Med J; 53:26-31
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Background] Friedland D, Hutchinson P. Classification of traumatic brain injury. Advances in Clinical Neuroscience and Rehabilitation. 27 Jul 2013.